CLINICAL TRIAL: NCT01421654
Title: Evaluation of Positive Airway Pressure (PAP) Feature to Improve Patient Adherence to Therapy
Brief Title: Evaluation of Acclimate Feature for Positive Airway Pressure (PAP) Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MA-03-11-01
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Results first posted 2013-03-07 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; Sleep Apnea; PAP; positive airway pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fixed Mode + Acclimate (Experimental): S9 Elite flow generator with Acclimate feature activated.
  Interventions: Device: S9 Elite with Acclimate
- Fixed Mode only (Active Comparator): S9 Elite Flow Generator with Fixed Mode only
  Interventions: Device: S9 Elite

INTERVENTIONS:
Device: S9 Elite with Acclimate — S9 Elite Flow Generator with Acclimate feature activated
  Arms: Fixed Mode + Acclimate
Device: S9 Elite — S9 Elite Flow Generator
  Arms: Fixed Mode only

SUMMARY:
The purpose of the study is to evaluate if using the Acclimate feature at the beginning of Positive Airway Pressure (PAP) therapy results in patients using their PAP therapy at least as long as they would standard therapy. Additionally, the Acclimate feature will be evaluated with regard to patient comfort, ease of acceptance of PAP therapy, leak events, and respiratory events.

DETAILED DESCRIPTION:
Acclimate has been designed as a comfort feature for patients starting PAP therapy. The feature allows acclimatization to the targeted positive airway pressure setting. Using the Acclimate feature, the pressure increases incrementally over a period of time. The feature can be only be used for a set period of time, afterwards which the device initiates the therapeutic session at the prescribed pressure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years of age.
* Recent diagnosis of moderate to severe OSA where fixed PAP is clinically indicated.
* Naïve to PAP therapy.

Exclusion Criteria:

* Patients requiring supplemental oxygen.
* Patients with a history of pneumothorax, pneumomediastinum, cavities or cysts in the lung.
* Previous surgery to the brain, middle or inner ear, pituitary gland or sinuses.
* Middle ear infection or perforated ear drum.
* Ongoing sinus infection/sinusitis.
* Clinically significant epistaxis.
* Predominant central sleep apneas in the subject's PSG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Plotkin, MD, Principal Investigator — Sleep Insights
Locations (1):
- Sleep Insights, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at one (1) clinical site in the US. The first subject was consented 06Sept2011 (Subject 01) and the last subject consented on 23Nov2011 (Subject 23).
Period: Overall Study
Arm/Group | Fixed Mode + Acclimate | Fixed Mode Only
Started | 11 | 9
Completed | 11 | 9 (10 subjects completed study, but 1 subject was found to not meet IEC at the end; data was not used.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed Mode + Acclimate | Fixed Mode Only | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 16
  >=65 years | 1 | 3 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 52.3 (11.2) | 58.5 (9.2) | 55.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Hours Used
Description: The number of hours that each group used the device will be compared between subjects using fixed pressure with the Acclimate mode and subjects using fixed pressure without the Acclimate mode.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Total Hours Used
Arm/Group | Fixed Mode + Acclimate | Fixed Mode Only
Number analyzed (Participants) | 11 | 9
Total Hours Used | 146.9 (62.9) | 141.9 (64.8)

ADVERSE EVENTS:
Arm/Group | Fixed Mode + Acclimate | Fixed Mode Only
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less